CLINICAL TRIAL: NCT02522416
Title: A Comparison of Two Devices for Measuring the Central Thickness of the Cornea Before and After Surgery (CECOT)
Acronym: CECOT
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JFO_2015_30
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Disorders, Refractive
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Central corneal thickness measurement

SUMMARY:
Corneal topography allows the measure of the radii of curvature and of the thickness of the cornea. It is essential for diagnosis in ophthalmology and allows to highlight corneal irregularities such as a keratoconus, or too thin corneas which are a contra-indication for laser refractive surgery.

Several types of corneal topographers are commercially available. Some as the Orbscan(r), operate by analyzing the image of the patterns of a Placido disk associated with a light slit, allowing the collection of thousands of points of the anterior and posterior surface of the cornea. More recent systems such as the Pentacam(r) are based on automatic rotary cameras which capture images of the whole anterior segment of the eye. The aim of this study is to compare two topographs, the Pentacam(r) and the Orbscan(r) and, more specifically, the central corneal pachymetry measurements measured pre- and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom a LASIK refractive surgery is planned

Exclusion Criteria:

* hyperopic patient
* another refractive surgery technique
* pregnant or lactating woman
* patient's opposition to participation in the study, according to the law on research into routine care
* patient under a measure of legal protection
* absence of affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for whom a LASIK refractive surgery at the Adolphe de Rothschild ophthalmologic foundation is planned
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Concordance of the Orbscan and Pentacam topographs, evaluated by the intra-class correlation coefficient, for the measure of the difference of the central thickness of the cornea before and after surgery. | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, Paris, France